CLINICAL TRIAL: NCT04343248
Title: A Randomized, Double-Blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Nitazoxanide (NTZ) for Post-Exposure Prophylaxis of COVID-19 and Other Viral Respiratory Illnesses in Elderly Residents of Long-Term Care Facilities (LTCF)
Brief Title: Trial to Evaluate the Efficacy and Safety of Nitazoxanide (NTZ) for Post-Exposure Prophylaxis of COVID-19 and Other Viral Respiratory Illnesses in Elderly Residents of Long-Term Care Facilities (LTCF)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study recruitment was halted prematurely as widespread vaccination of the study population made completion infeasible.
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RM08-3006
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: COVID-19; Viral Respiratory Illnesses
Keywords: COVID-19; Viral Respiratory Illnesses
MeSH Terms: conditions — COVID-19 | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Active Comparator): Two Nitazoxanide 300 mg tablets orally twice daily for 6 weeks
  Interventions: Drug: Nitazoxanide; Dietary Supplement: Vitamin Super B-Complex
- Placebo (Placebo Comparator): Two placebo tablets orally twice daily for 6 weeks
  Interventions: Drug: Placebo; Dietary Supplement: Vitamin Super B-Complex

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide 600 mg administered orally twice daily for six weeks
  Other Names: NTZ (nitazoxanide); NT-300
  Arms: Nitazoxanide
Drug: Placebo — Placebo administered orally twice daily for six weeks
  Arms: Placebo
Dietary Supplement: Vitamin Super B-Complex — Vitamin Super B-Complex administered orally twice daily to maintain the blind

SUMMARY:
Trial to evaluate the efficacy and safety of NTZ for post-exposure prophylaxis of COVID-19 and other VRIs in elderly LTCF residents.

DETAILED DESCRIPTION:
Multicenter, randomized, double-blind, placebo-controlled trial to evaluate the efficacy and safety of NTZ for post-exposure prophylaxis of COVID-19 and other VRIs in elderly LTCF residents.

ELIGIBILITY:
Inclusion Criteria:

* Male and female residents of LTCFs at least 55 years of age.
* Willing and able to provide written informed consent and comply with the requirements of the protocol.
* At least one symptomatic laboratory-confirmed COVID-19 illness identified among residents or staff of the LTCF within 10 days prior to randomization.

Exclusion Criteria:

* Alzheimer's disease, dementia, or other mental incapacity which precludes comprehension of the study requirements or symptom diary.
* Subjects expected to require hospitalization within the 8-week treatment and follow-up period.
* Subjects with a history of COVID-19 or known to have developed anti-SARS- CoV-2 antibodies.
* Subjects who experienced a previous episode of acute upper respiratory tract infection, otitis, bronchitis or sinusitis or received antibiotics for these conditions or antiviral therapy for influenza within two weeks prior to and including study day 1.
* Receipt of any dose of NTZ within 7 days prior to screening.
* Treatment with any investigational drug or vaccine within 30 days prior to screening or unwilling to avoid them during the course of the study.
* Known sensitivity to NTZ or any of the excipients comprising the study medication.
* Subjects unable to swallow oral tablets or capsules.
* Subjects taking medications considered to be major CYP2C8 substrates.
* Subjects who, in the judgment of the Investigator, will be unlikely to comply with the requirements of this protocol.

Ages: 55 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The Chappel Group Research, Kissimmee, Florida
  - Clinical Trial Specialists, Inc., Acworth, Georgia
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Centex Studies, Inc., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitazoxanide | Placebo
Started | 97 | 93
Completed | 81 | 78
Not Completed | 16 | 15
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 9 | 6
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population includes all subjects who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitazoxanide | Placebo | Total
Number analyzed (Participants) | 97 | 93 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (9.1) | 73 (10.0) | 74 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 75
  Male | 58 | 57 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 87 | 86 | 173
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 19 | 17 | 36
  White | 76 | 73 | 149
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Presence of anti-SARS-CoV-2 antibodies [Count of Participants; unit: Participants]
  Anti-SARS-CoV-2 antibodies present | 14 | 20 | 34
  Anti-SARS-CoV-2 antibodies absent | 78 | 65 | 143
  Unknown | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Laboratory-confirmed COVID-19
Description: The proportion of subjects with symptomatic laboratory-confirmed COVID-19 identified after start of treatment and before the end of the 6-week treatment period. NOTE: No statistical analyses were performed as enrollment was terminated early. See caveats and limitations.
Time Frame: up to 6 weeks
Population: The primary efficacy population consists of all subjects who received at least one dose of study medication and were negative for all respiratory viruses at Baseline. Proportions rounded to the nearest hundredth.
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 85 | 81
proportion of subjects | 0.01 | 0.00

2. Primary Outcome: Symptomatic Laboratory-confirmed VRI
Description: The proportion of subjects with symptomatic laboratory-confirmed VRI identified after the start of treatment and before the end of the 6-week treatment period. NOTE: No statistical analyses were performed as enrollment was terminated early. See caveats and limitations.
Time Frame: up to 6 weeks
Population: as for outcome 1
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 85 | 81
proportion of subjects | 0.01 | 0.00

3. Secondary Outcome: Hospitalization Due to COVID-19 or Complications Thereof
Description: Proportion of subjects hospitalized due to COVID-19 or complications thereof. NOTE: No statistical analyses were performed as enrollment was terminated early. See caveats and limitations
Time Frame: Up to 6 weeks
Population: The primary efficacy population consists of all subjects who received at least one dose of study medication and were negative for all respiratory viruses at Baseline.
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 85 | 81
proportion of subjects | 0.00 | 0.00

4. Secondary Outcome: Mortality Due to COVID-19 or Complications Thereof
Description: Proportion of subjects experiencing mortality due to COVID-19 or complications thereof. NOTE: No statistical analyses were performed as enrollment was terminated early. See caveats and limitations.
Time Frame: Up to 6 weeks
Population: as for outcome 3
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 85 | 81
proportion of subjects | 0.00 | 0.00

5. Secondary Outcome: Presence of Anti-SARS-CoV-2 at Weeks 6 or 8
Description: Proportion of subjects with anti-SARS-CoV-2 antibodies at Week 6 or 8 visits. NOTE: No statistical analyses were performed as enrollment was terminated early. See caveats and limitations.
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 85 | 81
proportion of subjects | 0.21 | 0.27

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Nitazoxanide | Placebo
All-Cause Mortality (participants affected / at risk) | 1/97 | 2/93
Serious Adverse Events (participants affected / at risk) | 10/97 | 8/93
Other Adverse Events (participants affected / at risk) | 8/97 | 9/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (N=97) | Placebo (N=93)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (N=97) | Placebo (N=93)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (7)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (6)

LIMITATIONS AND CAVEATS:
It was no longer possible to enroll eligible participants in the trial after vaccines were distributed to residents of long-term care facilities. Therefore, enrollment was terminated before the planned enrollment was completed. Study results are summarized descriptively, but no statistical analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT04343248/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT04343248/SAP_001.pdf